CLINICAL TRIAL: NCT06157086
Title: This is a Non-interventional, Prospective, Multicenter Study Conducted in France. The Primary Objective of This Study is to Describe the Quality of Life of MS Patients After Initiation of Treatment With Ofatumumab.
Brief Title: Assessment of the Quality of Life of Multiple Sclerosis Patients Treated With Ofatumumab in Real-life in France
Acronym: SEPROS
Status: Active, not recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: COMB157GFR06
Record Dates: First submitted 2023-11-27; First posted 2023-12-05 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Multiple Sclerosis (MS)
Keywords: MS; Multiple sclerosis; NIS; ofatumumab; Kesimpta; QoL; PRO
MeSH Terms: conditions — Multiple Sclerosis | interventions — ofatumumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ofatumumab: MS adult patients who initiated ofatumumab as per neurologist practice and regardless of the study protocol
  Interventions: Other: ofatumumab

INTERVENTIONS:
Other: ofatumumab — There is no treatment allocation. Participants with MS that initiated treatment with ofatumumabas per neurologist practice and regardless of the study protocol
  Other Names: KESIMPTA

SUMMARY:
SEPROS is a non-interventional study, based on primary data collection of MS adult patients who initiated ofatumumab as per neurologist practice and regardless of the study protocol.

DETAILED DESCRIPTION:
This is a non-interventional, prospective (primary data), multicenter study conducted in metropolitan France. The primary objective of this study is to describe the quality of life of MS patients after initiation of treatment with ofatumumab.

In order to form a representative sample of MS patients taking into account the terms of care in France, free or practicing neurologists in healthcare institutions (public or private) in different regions of France will be selected to participate in this study.

The study will enroll adult patients with MS who initiated ofatumumab according to the physician's advice and independently of the study. Patients will be followed from initiation of ofatumumab either until (i) 12 months (± 1month) after initiation of ofatumumab (End of Study), or until (ii) discontinuation of treatment with ofatumumab prior to the completion of the 12-month follow-up (early termination); whichever occurs first (end of study or early termination).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years of age or older
2. Patient with confirmed MS diagnosis
3. Patient initiating treatment with ofatumumab for the first time
4. Patient for which the decision to initiate treatment with ofatumumab was made by the doctor (investigator) in accordance with his/her usual practices independently of the study
5. Patient not opposed to participation in this study
6. Patient willing and able to complete patient questionnaires

Exclusion Criteria:

1. Patient treated with ofatumumab in the context of a clinical trial

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be adult patients with MS (women and men) who have initiated treatment with ofatumumab (Kesimpta ®).
Sampling Method: Non-Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2023-12-21 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Quality of life - MUSIQoL questionnaire | 12 months
  The primary objective of this non-interventional study is to describe the quality of life of adult patients with MS treated with ofatumumab in real life, in France, after 12 months of treatment with ofatumumab using the MUSIQoL Quality of Life Questionnaire.
  The MuSiQoL measures MS-specific quality of life. It comprises 31 items covering 9 domains (activities of daily living, psychological well-being, symptoms, relationships with friends, relationships with family, relationships with the healthcare system, sentimental and sexual life, coping, and rejection). Each item is scored on a 6-point Likert scale. The score on each dimension is obtained by computing the mean of the item scores for that dimension. All dimension scores are linearly transformed to a 0-100 scale. The global index score is computed as the mean of the dimension scores. Higher scores represent higher quality of life.

SECONDARY OUTCOMES:
Treatment satisfaction of patients treated with ofatumumab using TSQM 9 questionnaire | 12 months
  TSQM -9 is a self-questionnaire used to assess patient satisfaction with their treatment. It is a validated questionnaire and a good predictor of compliance. It explores 4 dimensions of satisfaction (efficacy, side effects, simplicity and overall satisfaction), through 9 questions. Responses are expressed on a 7-point Likert scale to precisely capture the patient's point of view. The responses to the items are aggregated; thus, each dimension is noted between 0 (extremely dissatisfied) and 100 (extremely satisfied).
Impact of MS on professional activity using the 6-item WPAI questionnaire | 12 months
  The WPAI measures absence, presence, decreased work productivity, and reduction in normal daily activities over the past 7 days. This self-questionnaire is non-specific for a disease and is developed in 6 questions. It works to calculate a health-related deterioration score, which combines the absence score and presence score. This deterioration score is rated between 0 and 1 where 1 corresponds to the maximum score, i.e. stopping work
Neurologist's decision criteria for initiating ofatumumab and patient involvement in the treatment choice | Baseline
  For each patient included in the study, neurologist's decision criteria for ofatumumab initiation will be collected (i.e., patient characteristics and poor prognosis factors or reasons for treatment switch if applicable) as well as the involvement of the patient in the choice of treatment (yes or no)
Clinical evolution of Multiple sclerosis - EDSS score | 12 months
  The Expanded Disability Status Scale (EDSS) is a method of quantifying disability in multiple sclerosis and monitoring changes in the level of disability over time. The EDSS scale ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability. Scoring is based on an examination by a neurologist.
Clinical evolution of Multiple sclerosis - Number of patients with relapses | Up to 12 months
  Number of patients with relapses and number of patients with hospitalizations related to the relapse
Number of patient adherent to ofatumumab from patient and practitioner perspectives | 12 months
  Number of patient adherent to ofatumumab from patient and practitioner perspectives to be collected
Ofatumumab discontinuation | 12 months
  Ofatumumab discontinuation by reason to be collected
Persistence on ofatumumab | Month 6, Month 12
  Patients still treated with ofatumumab at 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (46):
- France (46):
  - Novartis Investigative Site, Angers, France
  - Novartis Investigative Site, Paris, France
  - Novartis Investigative Site, Agen
  - Novartis Investigative Site, Altkirch
  - Novartis Investigative Site, Amiens
  - Novartis Investigative Site, Belfort
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Boulogne-sur-Mer
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Brunstatt Didenheim
  - Novartis Investigative Site, Cahors
  - Novartis Investigative Site, Chambéry
  - Novartis Investigative Site, Cherbourg Octeville
  - Novartis Investigative Site, Compiègne
  - Novartis Investigative Site, Contamine-sur-Arve
  - Novartis Investigative Site, Dax
  - Novartis Investigative Site, Gonesse
  - Novartis Investigative Site, Le Bouscat
  - Novartis Investigative Site, Le Coudray
  - Novartis Investigative Site, Lens
  - Novartis Investigative Site, Libourne
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Mantes-la-Jolie
  - Novartis Investigative Site, Marseille 01
  - Novartis Investigative Site, Meaux
  - Novartis Investigative Site, Metz-Tessy
  - Novartis Investigative Site, Mont-de-Marsan
  - Novartis Investigative Site, Montluçon
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Mulhouse
  - Novartis Investigative Site, Nîmes
  - Novartis Investigative Site, Orsay
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Poissy
  - Novartis Investigative Site, Quint-Fonsegrives
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Saverne
  - Novartis Investigative Site, Sélestat
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Tours
  - Novartis Investigative Site, Valence
  - Novartis Investigative Site, Vannes
  - Novartis Investigative Site, Villeurbanne

IPD SHARING:
Plan to Share IPD: No